CLINICAL TRIAL: NCT02049112
Title: Phase 4 Study Evaluating Efficacy, Safety and Acceptability of Treatment With a New Salivary Equivalent Compared to Two Moisturizing Mouth Sprays on the Improvement of Dry Mouth Symptoms and Oral Comfort in Patients With Xerostomia.
Brief Title: A New Oral salIvary equivAlent Compared to Two moisturizinG Mouth sprAys in Patients With xeRostomiA: NIAGARA Study
Acronym: NIAGARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unither Pharmaceuticals, France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UN/2011/001
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Xerostomia; Hyposalivation; Head and Neck Cancer; Sjögren Syndrome
Keywords: Cross-over; Salivary equivalent; Dry mouth; Medical device
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms; Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Salivary equivalent (Experimental): Single dose stick without any active substance
  Interventions: Device: Salivary equivalent
- Aequasyal (Sham Comparator): Multidose moisturizing oral spray without any active substance
  Interventions: Device: Aequasyal
- Biotene (Sham Comparator): Multidose moisturizing oral spray without any active substance
  Interventions: Device: Biotene

INTERVENTIONS:
Device: Salivary equivalent — 14-day treatment with salivary equivalent sticks
  Arms: Salivary equivalent
Device: Aequasyal — 14-day treatment with Aequasyal oral spray
  Arms: Aequasyal
Device: Biotene — 14-day treatment with Biotene oral spray
  Arms: Biotene

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy, safety and acceptability of our new oral salivary equivalent in the relief of signs and symptoms related to mouth dryness as compared to two distinct moisturizing currently marketed oral sprays (Aequasyal® & Biotene®) in patients with xerostomia due to chronic hyposalivation.

DETAILED DESCRIPTION:
National, multicentre, randomised, active controlled, crossover, open-label study using a 3-latin-square design.

200 evaluable patients have been recruited

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Aged 18 years or more,
* Clinical diagnosis of xerostomia by a severe reduction of salivation, as detected by patient's answers to few specific questions and measured by saliva volume at screening visit (test of saliva weight absorbed ≤ 0.1g/min)
* Any medical condition or treatment leading to a severe reduction of salivation related to either:
* Head and neck radiation therapy for cancer,
* Gougerot-Sjögren syndrome
* Medications known to induce xerostomia (psychotropic drugs, antihypertensive drugs)
* Dehydration, hypothyroidism, Parkinson's disease and/or diabetes mellitus
* Female patients must be post-menopausal or using a highly effective method for avoidance of pregnancy throughout the whole study duration, if childbearing potential.
* Able to understand and comply with the protocol procedures
* Willing and able to give their written informed consent
* Affiliated to the French National Health Insurance Program

Exclusion Criteria:

* Known hypersensitivity to one of the study products or to one of their components
* Any planned change in dosing of all known medications inducing mouth dryness
* Concomitant treatment for xerostomia symptoms without a scheduled 3 to 7-day withdrawal window
* Oral candidiasis as diagnosed by a microbiological test obtained from an unstimulated whole saliva sample until 3-week period from disease release
* Oral ulceration
* Alcohol (>2 glasses of wine/day), smoking (>10 cigarettes/day), caffeine and/or theine intake (>4 cups/day)
* Patients unable to fill out the questionnaires or to comply with the study protocol
* Dental infection
* Patients participating to another clinical trial at the time of the study entry or within 30 days prior to study enrolment
* Life-threatening condition at the time of the study
* Pregnant or lactating women and women of childbearing potential refusing to use adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-01; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Dry mouth discomfort | 14 days
  Patient evaluation through the completion of a self rated 100 mm long VAS score. Anchor points of the VAS score will be 0 representing the absence of any dry mouth symptoms and 100 representing the worst imaginable picture of dry mouth discomfort

SECONDARY OUTCOMES:
Mouth burning sensation | 14 days
  Patient evaluation through the completion of a self rated 100 mm long VAS score.
Speech difficulties | 14 days
  Patient evaluation through the completion of a self rated 100 mm long VAS score.
Chewing difficulties | 14 days
  Patient evaluation through the completion of a self rated 100 mm long VAS score.
Swallowing difficulties | 14 days
  Patient evaluation through the completion of a self rated 100 mm long VAS score.
Taste perversion | 14 days
  Patient evaluation through the completion of a self rated 100 mm long VAS score.
Medical device acceptability | 14 days
  Patient evaluation through the completion of a self rated 100 mm long VAS score.
Medical device safety assessment | 14 days
  Patient evaluation through the completion of a self rated 100 mm long VAS score.

CONTACTS AND LOCATIONS:
Overall Officials: Michel SALOM, Medical, Principal Investigator — Leopold Bellan Fundation
Locations (1):
- Leopold Bellan Private Hospital, Magnanville, France